CLINICAL TRIAL: NCT00629291
Title: Evaluation of Iron Overload in the Heart, Liver and Pancreas: Patients With Sickle β Thalassemia and Sickle Cell Anemia.
Brief Title: MRI Evaluation of Iron Overload in the Heart, Liver and Pancreas in Patients Receiving Multiple Blood Transfusions.
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Orly Goitein MD, Sheba medical center
Other Study IDs: SHEBA-07-4859-OG-CTIL
Record Dates: First submitted 2008-02-25; First posted 2008-03-05 (Estimated); Last update posted 2010-05-11 (Estimated); Status verified 2010-05

CONDITIONS: Iron Overload
Keywords: iron overload; Thalassemia; Anemia, Sickle Cell; Magnetic Resonance Imaging
MeSH Terms: conditions — Iron Overload; Thalassemia; Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — No biosepcimens retained
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Sickle cell anemia patients
- 2: Sickle cell β thalassemia

SUMMARY:
Sickle cell anemia and Sickle cell β thalassemia patients require multiple transfusions in order to avoid chronic anemia sequel. This regimen entails intrinsic deleterious effects, the majority of which are related to iron deposition in the reticuloendothelial system. Thus, iron is deposited in hepatic, myocardial and endocrine glands tissues. Tools available for iron load evaluation include serum ferrtin levels, liver biopsy and echocardiography, all are non specific.

The purpose of this work is to compare iron overload in the liver, heart and pancreas in Sickle cell anemia and Sickle cell β thalassemia patients using T2* MRI sequences.

DETAILED DESCRIPTION:
Sickle cell anemia and Sickle cell β thalassemia patients recieving multiple transfusions are exposed to the effects of iron deposition in the reticuloendothelial system, including cardiac muscle, liver and pancreas. Tools available for iron load evaluation include serum ferrtin levels, liver biopsy and echocardiography, all are non specific.

The purpose of this work is to compare iron overload in the liver, heart and pancreas in Sickle cell anemia and Sickle cell β thalassemia patients using T2* MRI sequences.

Patients and Methods: 27 Sickle cell anemia and 28 Sickle cell β thalassemia will undergo transthoracic echocardiography, cardiac MRI using T2* sequences and clinical and laboratory evaluation for iron overload including ferritin levels and oral glucose tolerance test

.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of Sickle cell anemia or Sickle cell β thalassemia having received multiple blood transfusions.

Exclusion Criteria:

* contraindication to MRI

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Sickle cell anemia and Sickle cell β thalassemia patients from dedicated outpatient hospital clinic.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
outcome measure: iron overload on T2* MRI in the heart , liver and pancreas. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Orly Goitein, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center , Imaging Dept, Tel Litwinsky, Tel Hashomer, Israel